CLINICAL TRIAL: NCT04111952
Title: The Efficacy and Safety of an Additional Vaginal Laser Treatment in Women Previously Treated With Laser for Gynecological Indications.
Brief Title: The Effect of Additional Laser Treatments.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0349-19-RMB
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Lax Vaginal Introitus
MeSH Terms: interventions — Lasers, Gas

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional laser treatment (Experimental): Women receiving a single laser treatment.
  Interventions: Device: CO2 laser
- Sham laser treatment (Sham Comparator): Women receiving sham laser treatment.
  Interventions: Device: Sham laser

INTERVENTIONS:
Device: CO2 laser — A single session of CO2 vaginal laser treatment
  Arms: Additional laser treatment
Device: Sham laser — A single session of sham laser treatment.
  Arms: Sham laser treatment

SUMMARY:
Women previously treated with vaginal CO2 laser will receive an additional treatment 6 months after cessation of previous laser treatment or a sham laser treatment. The efficacy and safety of the additional treatment will be assessed.

DETAILED DESCRIPTION:
The following study is intended to evaluate the efficacy and safety of an additional laser treatment for women previously treated for gynecological indications with laser treatments. Women will be randomized to one of 2 groups: 1. Study group-additional single laser treatment. 2. Control group-single sham laser treatment. All women will fill out validated questionnaires regarding sexual function, urinary stress incontinence and satisfaction after treatment. All women will be followed for an additional 6 months to evaluate the length of effect.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated with 3 laser treatments.
* Clear PAP test from the last 3 years.

Exclusion Criteria:

* Vaginal bleeding of unknown source.
* Vaginal surgery in the past 9 months.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 253 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2023-01-28 (Estimated)

PRIMARY OUTCOMES:
Length of effect | From the treatment session up to 6 months post-treatment
  The duration of symptom improvement.

SECONDARY OUTCOMES:
Female sexual function index | From the treatment session up to 6 months post-treatment
  Changes in the female sexual function index questionnaire score (range 0-35)
Sexual intercourse | From the treatment session up to 6 months post-treatment
  Improvement in the monthly rate of sexual intercourse
Urinary distress index | From the treatment session up to 6 months post-treatment
  Changes in the urinary distress index questionnaire score (range 0-15)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No